CLINICAL TRIAL: NCT06046560
Title: DRIVE Program: Diabetes Remote Intervention to improVe Use of Evidence-based Medications
Brief Title: Diabetes Remote Intervention to improVe Use of Evidence-based Medications
Acronym: DRIVE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Novo Nordisk A/S (Industry)
Responsible Party: Principal Investigator, Benjamin M. Scirica, MD, Associate Professor, Harvard Medical School, Brigham and Women's Hospital
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: 2020P003822
Record Dates: First submitted 2023-08-31; First posted 2023-09-21 (Actual); Results first posted 2024-10-23 (Actual); Last update posted 2024-10-23 (Actual); Status verified 2024-10

CONDITIONS: Cardiovascular Diseases; Diabetes
Keywords: Digital Health; Remote Care Delivery; Team-based Care Model
MeSH Terms: conditions — Cardiovascular Diseases; Diabetes Mellitus | interventions — Sodium-Glucose Transporter 2 Inhibitors

STUDY DESIGN:
Intervention Model Description: One group of patients, upon randomization, will immediately begin participation in a remote, pharmacist-driven clinic that will initiate and titrate medications according to a standardized medical algorithm. The comparator group will first receive curated patient education, an alert to providers, and provider education, and then after 2 months begin participation in the remote clinic.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Medication & Education-First (Active Comparator): Patient will immediately begin participation in a remote, pharmacist-driven heart failure clinic that will initiate and titrate medications according to a standardized medical algorithm.
  Interventions: Drug: SGLT2 inhibitor, GLP-1 RA
- Education-First (Experimental): Patient will first receive curated patient education, an alert to providers, and provider education, and then after 2 months begin participation in the remote clinic.
  Interventions: Drug: SGLT2 inhibitor, GLP-1 RA; Behavioral: Education-First

INTERVENTIONS:
Drug: SGLT2 inhibitor, GLP-1 RA — Immediate initiation of guideline-directed medical therapy. Will also immediately receive the same educational services provided in the "Education-First" intervention.
Behavioral: Education-First — For the first 2-months of their participation, patients in this arm will receive curated patient education, an alert to providers, provider education, and then after 2 months, be invited to participate in the remote clinic. The patient education would consist of curated video content and informational worksheets provided by email or secure patient messaging. Provider alerts would happen through notifying of a patient's eligibility for therapy.
  Arms: Education-First

SUMMARY:
A randomized remote, implementation trial in the Mass General Brigham network was performed on 200 patients with T2D at high CV or kidney risk. The study's primary objective was to create a remote diabetes management platform that improved the initiation and adherence to glucose-lowering medications with CV and kidney benefit and was evaluated by the primary outcome: increasing the proportion of patients with prescriptions for GDMT therapy by 6 months.

DETAILED DESCRIPTION:
A randomized remote, implementation trial in the Mass General Brigham network performed on 200 patients with T2D at high CV or kidney risk. Patients eligible for, but not prescribed, SGLT2i or GLP-1 RA were randomly assigned to 1) simultaneous patient education and medication initiation "simultaneous" arm or 2) 2-months of education followed by medication initiation "education-first" arm. A multi-disciplinary team provided education and prescribed GDMT using a treatment algorithm. The study's primary objective was to create a remote diabetes management platform that improved the initiation and adherence to glucose-lowering medications with CV and kidney benefit and was evaluated by the primary outcome: increasing the proportion of patients with prescriptions for GDMT therapy by 6 months. Secondary objectives included the primary outcome by randomization arm, prescribed therapy by 2 months, and patients taking prescribed therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 27 - 79 years at the time of agreeing to participate in the program
2. Presence of type 2 diabetes (treated with metformin unless intolerant, may also be treated with DPP4i, sulfonylurea, pioglitazone, and/or basal insulin)
3. HbA1c 6.5-8.9%; AND
4. At elevated cardiovascular and/or renal risk defined as any diagnosed ASCVD, estimated ASCVD risk >10%, congestive heart failure, non-alcoholic fatty liver disease, estimated glomerular filtration rate (eGFR) <60 mL/min/1.73m2, albuminuria above 300mg/g; and those aged 60 years or older with at least two of: active tobacco use, dyslipidemia (LDL-c above 160 mg/dL or 4.1 mmol/L, non-HDL-C above 190 mg/dL or 4.9 mmol/L, triglycerides above 175 mg/dL,) hypertension (2 systolic blood pressure values above 130 mmHg and/or 2 diastolic blood pressure values above 90 mmHg within 12 months,) or BMI above 30
5. Has seen a primary care provider within the Mass General Brigham network within the last year

Exclusion Criteria:

1. Type 1 diabetes
2. Currently or previously prescribed an SGLT2i or GLP1-RA
3. Taking any short-acting insulin
4. History of diabetic ketoacidosis
5. History of hypoglycemia requiring hospitalization
6. Frequent (more than two times in 1 week) episodes of symptomatic hypoglycemia with blood glucose <70 mg/dL
7. eGFR below 15 ml/min/m2
8. Mental incapacity, unwillingness, or language barriers precluding adequate understanding or cooperation, OR
9. Life expectancy less than 1 year or utilizing palliative care

Ages: 27 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2021-03-22 (Actual); Primary Completion 2023-07-25 (Actual); Study Completion 2023-07-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin M Scirica, MD MPH, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Background] Blood AJ, Chang LS, Colling C, Stern G, Gabovitch D, Feldman G, Adan A, Waterman F, Durden E, Hamersky C, Noone J, Aronson SJ, Liberatore P, Gaziano TA, Matta LS, Plutzky J, Cannon CP, Wexler DJ, Scirica BM. Methods, rationale, and design for a remote pharmacist and navigator-driven disease management program to improve guideline-directed medical therapy in patients with type 2 diabetes at elevated cardiovascular and/or kidney risk. Prim Care Diabetes. 2024 Apr;18(2):202-209. doi: 10.1016/j.pcd.2024.01.005. Epub 2024 Feb 1. PMID 38302335
- [Result] Blood AJ, Chang LS, Hassan S, Chasse J, Stern G, Gabovitch D, Zelle D, Colling C, Aronson SJ, Figueroa C, Collins E, Ruggiero R, Zacherle E, Noone J, Robar C, Plutzky J, Gaziano TA, Cannon CP, Wexler DJ, Scirica BM. Randomized Evaluation of a Remote Management Program to Improve Guideline-Directed Medical Therapy: The DRIVE Trial. Circulation. 2024 Jun 4;149(23):1802-1811. doi: 10.1161/CIRCULATIONAHA.124.069494. Epub 2024 Apr 7. PMID 38583146
- [Derived] Chang LS, Hassan S, Chasse J, Stern G, Gabovitch D, Zelle D, Colling C, Crossen J, Aronson SJ, Oates M, Figueroa C, Collins E, Ruggiero R, Plutzky J, Gaziano TA, Cannon CP, Wexler DJ, Scirica BM, Blood AJ. Safety of a remote disease management program to improve sodium-glucose cotransporter-2 inhibitors and glucagon-like peptide-1 receptor agonists prescribing in type 2 diabetes with elevated cardiovascular or kidney risk. Am Heart J. 2026 Jan 27:107359. doi: 10.1016/j.ahj.2026.107359. Online ahead of print. PMID 41610902

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Medication & Education-First | Education-First
Started | 116 | 84
Completed | 116 | 84
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Medication & Education-First | Education-First | Total
Number analyzed (Participants) | 116 | 84 | 200
Age, Continuous [Mean (Standard Deviation); unit: Years] | 66.6 (7.7) | 66.4 (7.5) | 66.5 (7.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42 | 31 | 73
  Male | 74 | 53 | 127
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 92 | 64 | 156
  Black | 14 | 10 | 24
  Asian | 6 | 4 | 10
  Other | 1 | 3 | 4
  Unknown | 2 | 2 | 4
  Declined | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Prescriptions of SGLT2i or GLP1-RA at Any Time
Description: Number of patients with prescriptions of SGLT2i or GLP1-RA at any time
Time Frame: Any time between 0-months (baseline) to 6-months following enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | Medication & Education-First | Education-First
Number analyzed (Participants) | 116 | 84
Participants | 81 | 47

2. Secondary Outcome: Number of Patients With Prescriptions of SGLT2i or GLP1-RA at 2-months
Description: Number of patients with prescriptions of SGLT2i or GLP1 RA at 2-months
Time Frame: 2-months following enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | Medication & Education-First | Education-First
Number analyzed (Participants) | 116 | 84
Participants | 62 | 7

3. Secondary Outcome: Number of Patients With Prescriptions of SGLT2i or GLP1-RA at 6-months
Description: Number of patients with prescriptions of SGLT2i or GLP1-RA at 6-months
Time Frame: At 6-months following enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | Medication & Education-First | Education-First
Number analyzed (Participants) | 116 | 84
Participants | 81 | 47

4. Secondary Outcome: Change in Short-form Patient Activation Measure (PAM)
Description: Change in Short-form Patient Activation Measure (PAM)
  The score is measured on a 0.0 - 4.0 point scale and indicates participants' relationships with and understanding of their health care. A higher value represents a better outcome. This measure indicates the change in participants' scores from the point of enrollment (0-months) to program completion (6-months).
  0.0 - 1.0 (Disengaged & Overwhelmed)
  1.1 - 2.0 (Becoming Aware But Still Struggling)
  2.1 - 3.0 (Taking Action & Gaining Control)
  3.1 - 4.0 (Maintaining Behaviors & Pushing Further)
Time Frame: From 0-months (baseline) to 6-months following enrollment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Medication & Education-First | Education-First
Number analyzed (Participants) | 65 | 46
score on a scale | 0.3 (0.9) | 0.0 (1.1)

5. Other Pre Specified Outcome: Change in Body Weight (kg)
Description: Change in body weight (kg)
Time Frame: From 0-months (baseline) to 6-months following enrollment
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Medication & Education-First | Education-First
Number analyzed (Participants) | 116 | 84
kg | -4.2 (5.0) | -2.5 (2.0)

6. Other Pre Specified Outcome: Change in Body Weight (%)
Description: Change in body weight (%)
Time Frame: From 0-months (baseline) to 6-months following enrollment
Measure: Mean (Standard Deviation); unit: % weight change
Arm/Group | Medication & Education-First | Education-First
Number analyzed (Participants) | 116 | 84
% weight change | -2.5 (5.3) | -2.0 (4.2)

7. Other Pre Specified Outcome: Change in Laboratory Measured HbA1c
Description: Change in laboratory measured HbA1c
Time Frame: From 0-months (baseline) to 6-months following enrollment
Measure: Mean (Standard Deviation); unit: % change in HbA1c
Arm/Group | Medication & Education-First | Education-First
Number analyzed (Participants) | 116 | 84
% change in HbA1c | -0.3 (0.8) | -0.3 (0.7)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected from Enrollment (Month 0) to the time of program completion. Participants are queued for graduation six months after enrollment or after initiating medication therapy and completing laboratory test and monitoring follow-up, whichever is later.
Description: Adverse events were only assessed for participants who started a study medication.
  Serious Adverse Events were only assessed if deemed "Possibly Related" or "Probably Related" to the study drug.
  The SAE definition also included urgent care visits.
  Systematic assessments were performed through phone call questionaires given to participants.
  Non-systematic assessment was performed for SAEs only at the end of the study through analysis of the electronic health records.
Arm/Group | Medication & Education-First | Education-First
All-Cause Mortality (participants affected / at risk) | 1/69 | 0/37
Serious Adverse Events (participants affected / at risk) | 2/69 | 0/37
Other Adverse Events (participants affected / at risk) | 36/69 | 14/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Medication & Education-First (N=69) | Education-First (N=37)
Urinary Tract Infection (Infections and infestations) | 1 | 0
Abdominal Pain (Gastrointestinal disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Medication & Education-First (N=69) | Education-First (N=37)
Genital Mycotic Infection (Infections and infestations) | 6 | 0
Urinary Tract Infection (Infections and infestations) | 2 | 0
Hypovolemia (Cardiac disorders) | 10 | 2 — Symptoms consistent with possible volume depletion
Hypoglycemia (Endocrine disorders) | 2 | 0 — Glucose <70 mg/dL
Severe hypoglycemia (Endocrine disorders) | 0 | 0 — Glucose <70 mg/dL and requiring assistance from another person
Nausea (Gastrointestinal disorders) | 7 | 6
Vomitting (Gastrointestinal disorders) | 2 | 1
Diarrhea (Gastrointestinal disorders) | 3 | 3
Abdominal pain (Gastrointestinal disorders) | 4 | 2

LIMITATIONS AND CAVEATS:
The PAM Survey (Secondary Outcome) completion rate experienced low participant engagement: 90 participants missing baseline, 171 missing 60 day, and 159 missing 180 day.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-11-09): https://cdn.clinicaltrials.gov/large-docs/60/NCT06046560/Prot_001.pdf
  • Statistical Analysis Plan (2023-11-16): https://cdn.clinicaltrials.gov/large-docs/60/NCT06046560/SAP_002.pdf